CLINICAL TRIAL: NCT07200921
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Trial on the Treatment of Hypertensive Intracerebral Hemorrhage With Naoxuekang Dropping Pills
Acronym: TCM-ICH
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: The Affiliated Hospital of Qingdao University (Other); Beijing Kangerfu Pharmaceutical Company Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024ZD0522203
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-08

CONDITIONS: Hypertensive Intracerebral Hemorrhage; Cerebral Small Vessel Diseases
Keywords: Hypertensive intracerebral hemorrhage; Cerebral small vessel disease; Naoxuekang Dropping Pills; Randomized controlled trial
MeSH Terms: conditions — Intracranial Hemorrhage, Hypertensive; Cerebral Small Vessel Diseases

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two parallel groups: the Naoxuekang group or the placebo control group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants in this group will receive Naoxuekang Dropping Pills (20 pills, three times daily) orally for 90 days, in addition to standardized guideline-based Western medical care.
  Interventions: Drug: Naoxuekang Dropping Pills
- Control Group (Placebo Comparator): Participants in this group will receive matched placebo pills (20 pills, three times daily) orally for 90 days, in addition to standardized guideline-based Western medical care.
  Interventions: Drug: Naoxuekang Matching Placebo

INTERVENTIONS:
Drug: Naoxuekang Dropping Pills — A traditional Chinese medicine. Each pill weighs 35mg. Dosage: 20 pills, three times daily, orally for 90 days.
  Arms: Experimental Group
Drug: Naoxuekang Matching Placebo — A placebo pill matched to Naoxuekang Dropping Pills in appearance, taste , size, and packaging. Dosage: 20 pills, three times daily, orally for 90 days.
  Arms: Control Group

SUMMARY:
This study aims to evaluate the effectiveness and safety of a Chinese medicine-based intervention combined with standard medicine, in reducing composite vascular events in patients with hypertensive intracerebral hemorrhage (HICH).This is a multicenter, randomized, double-blind, placebo-controlled trial. A total of 1950 participants with HICH within 7 days of onset, accompanied by imaging evidence of cerebral small vessel disease, will be enrolled.Participants will be randomly assigned to receive eitherNaoxuekang Dropping Pills or matching placebo for 90 days, in addition to guideline-based standard care.The primary outcome is the incidence of composite vascular events (including ischemic stroke, hemorrhagic stroke, myocardial infarction, vascular death, deep vein thrombosis, and pulmonary embolism) within 1 year.Secondary outcomes include vascular events within 90 days, neurological function (mRS), and cognitive function (MMSE, MoCA) at 90 days and 1 year.Safety will be monitored through adverse event reporting.The results will provide evidence for optimizing secondary prevention strategies in HICH patients.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the diagnostic criteria for hypertensive intracerebral hemorrhage.
2. Able to cooperate with a head MRI examination and has imaging manifestations of cerebral small vessel disease (CSVD) (Staals total CSVD burden score ≥ 1).
3. Supratentorial hemorrhage (volume ≤ 30ml) or infratentorial hemorrhage (volume ≤ 10ml).
4. Within 7 days of symptom onset.
5. NIHSS score ≤ 25.
6. GCS score ≥ 8.
7. Age between 18 and 80 years (inclusive).
8. Any gender

Exclusion Criteria:

1. Primary intraventricular hemorrhage.
2. Spontaneous intracerebral hemorrhage due to other causes or secondary intracerebral hemorrhage (e.g., from trauma, vascular malformations, coagulation disorders, hematological diseases, systemic diseases, or tumors).
3. Planned surgical intervention (including craniotomy for hematoma evacuation, minimally invasive hematoma removal, or ventricular puncture).
4. Patients with active peptic ulcer, bleeding, or other clear tendency for rebleeding.
5. Patients with severe hepatic or renal dysfunction (Severe hepatic dysfunction: ALT or AST > 3 times the upper limit of normal; Severe renal dysfunction: Serum creatinine > 2 times the upper limit of normal).
6. Suffering from other life-threatening severe diseases with an expected survival time of less than 1 year.
7. Known allergy to any component of the study drug.
8. Pregnant women, women planning pregnancy, or lactating women.
9. Participating in another interventional clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1950 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Composite Vascular Events | Within 1 year after the onset of intracerebral hemorrhage.
  Composite vascular events within one year of onset, including arterial vascular events (ischemic stroke, hemorrhagic stroke, myocardial infarction, vascular death) and venous vascular events (lower extremity venous thrombosis, pulmonary embolism).

CONTACTS AND LOCATIONS:
Overall Officials: Qian Zhang, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided